CLINICAL TRIAL: NCT07173608
Title: Transforming Adolescent Perception and Mental Health Through Meditation and Cognitive Reappraisal A Mixed Method Study
Acronym: THRIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Principal Investigator, Sepideh Hariri, Instructor in Anesthesia at Harvard Medical School, Program Manager at Department of Anesthesia, Beth Israel Deaconess Medical Center, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025P000560
Record Dates: First submitted 2025-08-21; First posted 2025-09-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Meditation; Cognitive Reappraisal; Emotional Regulation
Keywords: meditation; Inner Engineering; Shambhavi Mahamudra Kriya; EEG; Functional MRI; MRI; Cognition; Mindfulness; Mental Health; Adolescent
MeSH Terms: conditions — Emotional Regulation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a Randomized Controlled Trial with 48 intervention and 48 control adolescents (aged 15-18) to be followed up for 3 months. Subjects will be recruited from meditation-Naïve healthy individuals. The intervention group will complete the intervention training and learn a 21-minute meditation to practice daily. Various outcomes related to mental health and perception will be collected over a period of 3 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention participants will take the Inner Engineering program and are asked to practice meditation daily for the duration of the study.
  Interventions: Behavioral: Inner Engineering Program
- Control (No Intervention): Control participants will be asked to continue their daily routine

INTERVENTIONS:
Behavioral: Inner Engineering Program — The intervention is a comprehensive secular training called Inner Engineering (IE), offered by the international non-profit Isha Foundation. This program combines cognitive reappraisal and emotion regulation strategies, breath-based meditation and simple yoga practices. The training provides precise, step by step and easy to follow instructions on how to perform the practices. No previous experience of yoga and meditation is required. By fostering health, exuberance and awareness, one can "engineer their inner climate the way they want it" to lead a joyful, fulfilling life. Previous research shows improved wellbeing, mindfulness, joy, sleep, relationships, psychological capital, and work engagement, compassion, and parent-child relationships. Evidence suggest it may promote enhanced Heart Rate Variability and Sympathovagal balance.
  Arms: Intervention

SUMMARY:
This study will evaluate how a comprehensive meditation-based program, Inner Engineering, supports teens ages 15-18 in becoming more joyful, focused, resilient, and better equipped to manage stress and thrive. Through this study, researchers will examine whether practices like meditation, yoga, and cognitive reframing can help adolescents view and respond to challenges with greater clarity and balance. The study will assess mental and physical impacts through self-report, physiological, and neuroimaging methods.

DETAILED DESCRIPTION:
Adolescence is a critical developmental period marked by heightened vulnerability to mental health challenges and increased neuroplasticity, making it an ideal window for preventive interventions. This mixed-method randomized controlled trial (RCT) evaluates the efficacy of a secular, multimodal contemplative program-Inner Engineering-in enhancing psychological wellbeing, cognitive flexibility, and physiological balance among adolescents aged 15-18. Participants (N=96) will be randomized to either the intervention or a meditation-naïve control group.

The intervention training integrates cognitive reappraisal, breath-based meditation, and yoga-based postures, followed by daily practice. Assessments will occur at baseline, 6 weeks, and 12 weeks, and will include self-report questionnaires, behavioral tasks, EEG, fMRI, wearable physiological monitoring (including heartrate, sleep, respiration), and blood-based biomarkers of inflammation and neuroplasticity. Qualitative interviews will provide additional insight into the lived experiences of intervention participants.

The intervention aims to enabling more adaptive, inclusive, and empowered ways of perceiving external situations and internal states.

This is the first comprehensive RCT to investigate the multidimensional impact of an integrated contemplative program on the developing adolescent mental health, physiological and neural outcomes and perception . Findings may support scalable, evidence-based contemplative education tools to promote clarity, resilience, and expanded perception in youth.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between15-18 years of age
* Ability to understand study instructions and provide informed consent/assent. (parental consent for minors)
* Access to internet and a device to complete online study activities
* Currently residing in the United States
* Willing and able to travel to the hospital location in Boston for study procedures.

Exclusion Criteria:

* Non-English speaking (Justification: the intervention and assessment instruments are not validated in a sufficient range of languages, and the research team lacks polylingual capabilities or the financial resources to hire interpreters for the duration of all proposed assessments.)
* Practicing meditation regularly in the past 6 months (4 or more times per week for 4 weeks or more in the past 6 months)
* History of psychiatric illness such as severe anxiety, severe depression, posttraumatic stress disorder (PTSD), Schizophrenia or bipolar disorder
* Current use of cognition enhancing drugs
* Current management for chronic pain
* History (within past 5 years) of seizure, brain surgery or any condition causing cognitive decline.
* Active history (within the last 5 years) of alcohol or drug abuse.
* Current pregnancy or planning to become pregnant in the next 6 months
* Currently enrolled in another interventional study that could impact the primary outcome, as determined by the PI
* Significant visual impairment
* Subject has previously learned the intervention.
* Subject has contraindications for MRI (Detailed in the eligibility screening questions)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Emotional Wellbeing | Measured at Baseline, 6 weeks and 3 months
  the PERMA profiler, (15 items) designed to measure Seligman's five pillars of wellbeing (PERMA is the acronym developed from the first letter of these five pillars): Positive emotions, Relationships, Engagement, Meaning, and Accomplishment. It shows good reliability among adolescents and good construct validity. The total PERMA-Profiler score is the average of all the factor scores, which can range from 0 to 10, with higher scores indicating greater mental wellbeing.

SECONDARY OUTCOMES:
Depression, Anxiety and Stress | Measured at Baseline, 6 weeks and 3 months
  The Depression Anxiety Stress Scales - Youth version (DASS-Y) (21-items) is designed to measure general psychological distress and negative emotional states. The scale shows good construct validity as it has strong associations with physiological hyperarousal and excessive worrying. The total score can range from 0 to 63, with higher scores indicating a greater presence of psychological distress and negative emotional states.
Cognitive Flexibility | Measured at Baseline, 6 weeks and 3 months
  Cognitive Flexibility assessed via the Cognitive Flexibility Inventory (CFI) (20 items) to monitor how individuals challenge maladaptive thoughts. CFI has excellent internal consistency, and high 7-week test- retest reliability. The total score can range between 20 and 140, where higher scores indicate more cognitive flexibility.
Cognitive Emotion Regulation | Measured at Baseline, 6 weeks and 3 months
  Regulation strategies assessed via Cognitive Emotion Regulation questionnaire -short 18-item version (CERQ-short) with nine subscales (Self-blame, Other-blame, Rumination, Catastrophizing, Positive refocusing, Planning, Positive reappraisal, Putting into perspective and Acceptance). The reliability of the scales was found to be acceptably high among adolescents. The total possible score can range between 18 and 90, with higher scores indicating a greater use of cognitive emotion regulation strategies.
Personality Trait | Will be measured at Baseline, 6 weeks and 3 months
  Openness assessed via The Big Five Personality Trait Short Questionnaire (BFPTSQ) (10 item) assessing Openness, Extraversion, Agreeableness, Conscientiousness, and Emotional Stability. It has good reliability and convergent validity. Each personality type will get a score range of 1 to 7, with higher scores indicating the presence of that personality type.
Mindfulness | Will be measured at Baseline, 6 weeks and 3 months
  Mindful awareness is assessed via the Five Facet Mindfulness Questionnaire (FFMQ) with 5 subscales: Observing, Describing, Acting with Awareness, Nonjudgement and Non-reactivity. FFMQ-A-SF consists of 25 items (5 per facet) especially developed for adolescents. It shows good internal consistency and high construct validity. The total FFMQ score ranges from 39 to 195, with higher scores indicating greater mindfulness.
Sleep Quality | Will be measured at Baseline, 6 weeks and 3 months
  Pittsburg Sleep Quality Index (PSQI) is a widely used, validated self-report questionnaire that assesses sleep quality and disturbances over a 1-month interval. It consists of 19 items that generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. These components are summed to produce a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality.

OTHER OUTCOMES:
Qualitative Assessment | Will be measured at 6 weeks
  Open ended phenomenological interviews (individual and focus group) will be conducted to understand the intervention group's lived experience of practicing the intervention, and its impact on Perception Box and wellbeing. All these interviews will be conducted virtually via zoom, after they have learnt the intervention and been practicing it for at least 4 weeks. The interviews will last for about 30-45 minutes each.
Resting Heart Rate | Will be measured at Baseline, 6 weeks and 3 months
  Fitbit Wearable Smart Watches will be worn for 7 consecutive days use to assess resting heart rate.
Heart Rate Variability | Will be measured at Baseline, 6 weeks and 3 months
  Fitbit Wearable Smart Watches will be worn for 7 consecutive days to assess changes in heart rate, called heart rate variability. a higher value of heart rate variability indicates better cardiovascular health.
Blood Proteins | Measured at Baseline and 3 months
  SOMAScan Proteomics technology will be used to assess 11,000 proteins in blood plasma to observe any differences between the intervention and control groups.
Change in Frontal Midline Theta Power | Measured at Baseline and 3 months
  Frontal Midline Theta Power is obtained from an average of electrodes around the midline in a standard EEG cap and has been proposed as a correlate of meditation success in previous studies. Increased value suggests increased control over the brain's default mode network, suggesting more successful meditation experience.
  Time Frame: Measured at Baseline and 6 months
Change in Gamma Slope Index (GSI) | Measured at Baseline and 3 months
  GSI is an indicator of the Excitation-Inhibition (E-I) balance in the brain and is computed from the power spectral density slope of oscillatory activity in the brain, taking the low-gamma (40-60Hz) band slope of the Power Spectral Density, and is steeper (more negative) when the E-I balance is tipped towards more inhibition. A higher negative value suggests shift of the brain's excitation/inhibition balance toward more inhibition, indicating a calmer brain.
Changes in Brain Regional Volume | Measured at Baseline and 3 months
  Brain regional volume (mm^3) will be assessed using MRI. Brain regional volume is the volume of brain matter. Group-wise comparisons will be made between the intervention group and control. A positive difference between the intervention and control groups indicates greater brain volume.
Change in Brain Connectivity | Measured at Baseline and 3 months
  fMRI is an indirect measure of brain activity based on blood oxygen level dependent (BOLD) signals. Based on BOLD signals, functional connectivity will be assessed. Functional connectivity between two regions will be assessed for both the intervention and control group. A t-statistics value will be calculated based on the differences in signal intensities between the two groups. A more positive t-statistic indicates greater brain connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Sepideh Hariri, PhD, Principal Investigator — Beth Israel Deaconess Medical Centre, Boston, Massachusetts 02115

REFERENCES:
- [Background] Fox KC, Dixon ML, Nijeboer S, Girn M, Floman JL, Lifshitz M, Ellamil M, Sedlmeier P, Christoff K. Functional neuroanatomy of meditation: A review and meta-analysis of 78 functional neuroimaging investigations. Neurosci Biobehav Rev. 2016 Jun;65:208-28. doi: 10.1016/j.neubiorev.2016.03.021. Epub 2016 Mar 28. PMID 27032724
- [Background] Rodrigues E, Lima D, Barbosa P, Gonzaga K, Guerra RO, Pimentel M, Barbosa H, Maciel A. HRV Monitoring Using Commercial Wearable Devices as a Health Indicator for Older Persons during the Pandemic. Sensors (Basel). 2022 Mar 4;22(5):2001. doi: 10.3390/s22052001. PMID 35271148
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cortazar N, Calvete E, Fernandez-Gonzalez L, Orue I. Development of a Short Form of the Five Facet Mindfulness Questionnaire-Adolescents for Children and Adolescents. J Pers Assess. 2020 Sep-Oct;102(5):641-652. doi: 10.1080/00223891.2019.1616206. Epub 2019 Jun 5. PMID 31166802
- [Background] Baer RA, Carmody J, Hunsinger M. Weekly change in mindfulness and perceived stress in a mindfulness-based stress reduction program. J Clin Psychol. 2012 Jul;68(7):755-65. doi: 10.1002/jclp.21865. Epub 2012 May 23. PMID 22623334
- [Background] Morizot J. Construct validity of adolescents' self-reported big five personality traits: importance of conceptual breadth and initial validation of a short measure. Assessment. 2014 Oct;21(5):580-606. doi: 10.1177/1073191114524015. Epub 2014 Mar 11. PMID 24619971
- [Background] Saetren SS, Hegelstad WTV, Tjora T, Hafstad GS, Augusti EM. Validation of the short version of Cognitive Emotion Regulation Questionnaire for adolescents in Norway. Scand J Public Health. 2025 Feb;53(1):32-40. doi: 10.1177/14034948231225616. Epub 2024 Feb 1. PMID 38303505
- [Background] Szabo M, Lovibond PF. Development and Psychometric Properties of the DASS-Youth (DASS-Y): An Extension of the Depression Anxiety Stress Scales (DASS) to Adolescents and Children. Front Psychol. 2022 Apr 14;13:766890. doi: 10.3389/fpsyg.2022.766890. eCollection 2022. PMID 35496218
- [Background] Fernandes I, Zanini DS, Peixoto EM. PERMA-Profiler for adolescents: validity evidence based on internal structure and related constructs. Front Psychol. 2024 Jul 12;15:1415084. doi: 10.3389/fpsyg.2024.1415084. eCollection 2024. PMID 39070577
- [Background] Bruining H, Hardstone R, Juarez-Martinez EL, Sprengers J, Avramiea AE, Simpraga S, Houtman SJ, Poil SS, Dallares E, Palva S, Oranje B, Matias Palva J, Mansvelder HD, Linkenkaer-Hansen K. Measurement of excitation-inhibition ratio in autism spectrum disorder using critical brain dynamics. Sci Rep. 2020 Jun 8;10(1):9195. doi: 10.1038/s41598-020-65500-4. PMID 32513931
- [Background] Orekhova EV, Stroganova TA, Schneiderman JF, Lundstrom S, Riaz B, Sarovic D, Sysoeva OV, Brant G, Gillberg C, Hadjikhani N. Neural gain control measured through cortical gamma oscillations is associated with sensory sensitivity. Hum Brain Mapp. 2019 Apr 1;40(5):1583-1593. doi: 10.1002/hbm.24469. Epub 2018 Dec 13. PMID 30549144
- [Background] Gao R, Peterson EJ, Voytek B. Inferring synaptic excitation/inhibition balance from field potentials. Neuroimage. 2017 Sep;158:70-78. doi: 10.1016/j.neuroimage.2017.06.078. Epub 2017 Jul 1. PMID 28676297
- [Background] Brandmeyer T, Delorme A. Closed-Loop Frontal Midlinetheta Neurofeedback: A Novel Approach for Training Focused-Attention Meditation. Front Hum Neurosci. 2020 Jun 30;14:246. doi: 10.3389/fnhum.2020.00246. eCollection 2020. PMID 32714171
- [Background] Brandmeyer T, Delorme A. Reduced mind wandering in experienced meditators and associated EEG correlates. Exp Brain Res. 2018 Sep;236(9):2519-2528. doi: 10.1007/s00221-016-4811-5. Epub 2016 Nov 4. PMID 27815577
- [Background] van Loon AWG, Creemers HE, Okorn A, Vogelaar S, Miers AC, Saab N, Westenberg PM, Asscher JJ. The effects of school-based interventions on physiological stress in adolescents: A meta-analysis. Stress Health. 2022 Apr;38(2):187-209. doi: 10.1002/smi.3081. Epub 2021 Jul 26. PMID 34275188
- [Background] Pascoe MC, Thompson DR, Jenkins ZM, Ski CF. Mindfulness mediates the physiological markers of stress: Systematic review and meta-analysis. J Psychiatr Res. 2017 Dec;95:156-178. doi: 10.1016/j.jpsychires.2017.08.004. Epub 2017 Aug 23. PMID 28863392
- [Background] Chen W, Zhong Q, Chen H, Chen S. Heart rate variability in children and adolescents with major depressive disorder: A systematic review and meta-analysis. J Affect Disord. 2023 Aug 15;335:204-215. doi: 10.1016/j.jad.2023.05.022. Epub 2023 May 11. PMID 37178829
- [Background] Baumeister-Lingens L, Rothe R, Wolff L, Gerlach AL, Koenig J, Sigrist C. Vagally-mediated heart rate variability and depression in children and adolescents - A meta-analytic update. J Affect Disord. 2023 Oct 15;339:237-255. doi: 10.1016/j.jad.2023.07.027. Epub 2023 Jul 10. PMID 37437729
- [Background] Sharma A, Newberg AB. Mind-Body Practices and the Adolescent Brain: Clinical Neuroimaging Studies. Adolesc Psychiatry (Hilversum). 2015;5(2):116-124. doi: 10.2174/2210676605666150311223728. PMID 27347478
- [Background] Young KS, Sandman CF, Craske MG. Positive and Negative Emotion Regulation in Adolescence: Links to Anxiety and Depression. Brain Sci. 2019 Mar 29;9(4):76. doi: 10.3390/brainsci9040076. PMID 30934877
- [Background] Lichenstein SD, Verstynen T, Forbes EE. Adolescent brain development and depression: A case for the importance of connectivity of the anterior cingulate cortex. Neurosci Biobehav Rev. 2016 Nov;70:271-287. doi: 10.1016/j.neubiorev.2016.07.024. Epub 2016 Jul 25. PMID 27461914
- [Background] Creswell JD, Irwin MR, Burklund LJ, Lieberman MD, Arevalo JM, Ma J, Breen EC, Cole SW. Mindfulness-Based Stress Reduction training reduces loneliness and pro-inflammatory gene expression in older adults: a small randomized controlled trial. Brain Behav Immun. 2012 Oct;26(7):1095-101. doi: 10.1016/j.bbi.2012.07.006. Epub 2012 Jul 20. PMID 22820409
- [Background] Alvarez-Lopez MJ, Conklin QA, Cosin-Tomas M, Shields GS, King BG, Zanesco AP, Kaliman P, Saron CD. Changes in the expression of inflammatory and epigenetic-modulatory genes after an intensive meditation retreat. Compr Psychoneuroendocrinol. 2022 Jun 23;11:100152. doi: 10.1016/j.cpnec.2022.100152. eCollection 2022 Aug. PMID 35818436
- [Background] Kuhlman KR, Chiang JJ, Horn S, Bower JE. Developmental psychoneuroendocrine and psychoneuroimmune pathways from childhood adversity to disease. Neurosci Biobehav Rev. 2017 Sep;80:166-184. doi: 10.1016/j.neubiorev.2017.05.020. Epub 2017 May 31. PMID 28577879
- [Background] Danese A, Caspi A, Williams B, Ambler A, Sugden K, Mika J, Werts H, Freeman J, Pariante CM, Moffitt TE, Arseneault L. Biological embedding of stress through inflammation processes in childhood. Mol Psychiatry. 2011 Mar;16(3):244-6. doi: 10.1038/mp.2010.5. Epub 2010 Feb 16. No abstract available. PMID 20157309
- [Background] Gard T, Holzel BK, Lazar SW. The potential effects of meditation on age-related cognitive decline: a systematic review. Ann N Y Acad Sci. 2014 Jan;1307:89-103. doi: 10.1111/nyas.12348. PMID 24571182
- [Background] Chiesa A, Serretti A, Jakobsen JC. Mindfulness: top-down or bottom-up emotion regulation strategy? Clin Psychol Rev. 2013 Feb;33(1):82-96. doi: 10.1016/j.cpr.2012.10.006. Epub 2012 Oct 23. PMID 23142788
- [Background] Jafari N, Manvelian A, Mohamed E, Rayapuraju A, Orui H, Alkuhaimi S, Reed PU, Subramaniam B. Inner engineering is associated with perceived improvements in relationship quality, interpersonal connections, and interpersonal compassion. Front Psychol. 2024 Dec 23;15:1454293. doi: 10.3389/fpsyg.2024.1454293. eCollection 2024. PMID 39764085
- [Background] Hagen I, Skjelstad S, Nayar US. Promoting mental health and wellbeing in schools: the impact of yoga on young people's relaxation and stress levels. Front Psychol. 2023 May 17;14:1083028. doi: 10.3389/fpsyg.2023.1083028. eCollection 2023. PMID 37265958
- [Background] Muralikrishnan K, Balakrishnan B, Balasubramanian K, Visnegarawla F. Measurement of the effect of Isha Yoga on cardiac autonomic nervous system using short-term heart rate variability. J Ayurveda Integr Med. 2012 Apr;3(2):91-6. doi: 10.4103/0975-9476.96528. PMID 22707866
- [Background] Peterson CT, Bauer SM, Chopra D, Mills PJ, Maturi RK. Effects of Shambhavi Mahamudra Kriya, a Multicomponent Breath-Based Yogic Practice ( Pranayama), on Perceived Stress and General Well-Being. J Evid Based Complementary Altern Med. 2017 Oct;22(4):788-797. doi: 10.1177/2156587217730934. Epub 2017 Sep 22. PMID 29228793
- [Background] Chang TFH, Ramburn TT, Pundir S, Purandare P, Subramaniam B. The Effect of the Inner Engineering Online Program as a Positive Intervention on Subjective Well-Being and Positive Work Outcomes. J Integr Complement Med. 2022 Mar;28(3):278-282. doi: 10.1089/jicm.2021.0180. Epub 2022 Jan 31. PMID 35100026
- [Background] Immordino-Yang, M. H., Darling-Hammond, L., & Krone, C. R. (2019). Nurturing Nature: How Brain Development Is Inherently Social and Emotional, and What This Means for Education. Educational Psychologist, 54(3), 185-204. https://doi.org/10.1080/00461520.2019.1633924
- See also: Social and Emotional Learning Programs for Adolescents. Future of Children, — https://eric.ed.gov/?id=EJ1145078
- See also: The descriptive phenomenological method in psychology: A modified Husserlian approach — https://catalog.nlm.nih.gov/discovery/fulldisplay/alma9915137153406676/01NLM_INST:01NLM_INST